CLINICAL TRIAL: NCT05023915
Title: High-dose Dexamethasone Plus Diammonium Glycyrrhizinate Enteric-coated Capsule Versus High-dose Dexamethasone in Treatment-naive Primary Immune Thrombocytopenia (ITP): a Multicentre, Randomised, Open-label Trial
Brief Title: A Multicenter Randomized Open-label Study of Diammonium Glycyrrhizinate Enteric-coated Capsule Plus DXM Versus DXM in Treatment of ITP
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITP-Diammonium Glycyrrhizinate
Record Dates: First submitted 2021-08-21; First posted 2021-08-27 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Immune Thrombocytopenia
Keywords: Dexamethasone; Diammonium Glycyrrhizinate Enteric-coated Capsule
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- diammonium glycyrrhizinate enteric-coated capsule + high-dose dexamethasone (Active Comparator): Diammonium glycyrrhizinate enteric-coated capsule orally at a dose of 150mg tid for 1 month, combining with dexamethasone (given orally at a dose of 40 mg qd for 4 days). Patients who do not respond to the treatment may receive another cycle of high-dose dexamethasone therapy with an interval of 10 days.
  Interventions: Drug: dexamethasone; Drug: diammonium glycyrrhizinate enteric-coated capsule
- High-dose dexamethasone (Active Comparator): Dexamethasone orally at a dose of 40 mg qd for 4 days. Patients who do not respond to the treatment may receive another cycle of high-dose dexamethasone therapy with an interval of 10 days.
  Interventions: Drug: dexamethasone

INTERVENTIONS:
Drug: dexamethasone — 40 mg qd for 4 days
Drug: diammonium glycyrrhizinate enteric-coated capsule — 150mg tid for 1 month
  Arms: diammonium glycyrrhizinate enteric-coated capsule + high-dose dexamethasone

SUMMARY:
The project was undertaking by Qilu Hospital of Shandong University in China. In order to report the efficacy and safety of diammonium glycyrrhizinate enteric-coated capsule plus high-dose dexamethasone for the treatment of adults with newly-diagnosed primary immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
The investigators anticipate to undertaking a parallel group, randomised controlled trial of 106 ITP patients. One part of the participants are randomly selected to receive diammonium glycyrrhizinate enteric-coated capsule orally at a dose of 150mg tid for 1 month), combining with dexamethasone (given orally at a dose of 40 mg qd for 4 days). The others are selected to receive high-dose of dexamethasone alone. Patients who do not respond to the treatment may receive another cycle of high-dose dexamethasone therapy with an interval of 10 days. Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study. The purpose of this study is to report the efficacy and safety of diammonium glycyrrhizinate enteric-coated capsule combining with high-dose dexamethasone therapy for the treatment of ITP.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for immune thrombocytopenia;
* Untreated hospitalized patients or patients from the clinic, may be male or female, between the ages of 18~ 80 years;
* To show a platelet count <30 * 10^9/L, or with bleeding manifestations, or both;
* Willing and able to sign written informed consent
* ITP patients with hepatitis virus infection or ITP patients with abnormal liver function at the time of enrollment, i.e., ITP patients with indications for diammonium glycyrrhizinate enteric-coated capsule, should be separately stratified.

Exclusion Criteria:

* secondary thrombocytopenia;
* severe immune-deficiency;
* active or previous malignancy;
* HIV virus infection, tuberculosis, or other active infection (sepsis, pneumonia, or abscess);
* pregnancy or lactation;
* diabetes;
* hypertension;
* cardiovascular diseases;
* severe kidney function impairment;
* psychosis;
* osteoporosis;
* inflammatory bowel disease or gastric disease;
* arterial or venous thromboembolism within the 6 months before screening or patients who required anticoagulant treatment;
* an organ or haematopoietic stem-cell transplantation;
* neutrophil count of less than 1500 cells per mm³;
* glycosylated haemoglobin less than 8%;
* partial thromboplastin time 1∙5 times or less the upper limit of normal (ULN); •clinical electrocardiogram changes;
* history of primary immunodeficiency;
* neoplastic disease within the past 5 years;
* corrected QT interval greater than 450 ms for men and greater than 470 ms for women;
* substance misuse within the previous 12 months;
* people who could not adhere to the protocol or were planning to have a surgical procedure in 6 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2021-08-21 (Actual); Primary Completion 2021-08-21 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
14-day initial overall response to ITP treatments | 14 days after treatment started
  Complete response was defined as a platelet count of 100×10⁹ cells per L or higher and an absence of bleeding. Partial response was defined as a platelet count of 30×10⁹ cells per L or higher, but less than 100×10⁹ cells per L, and at least a doubling of the baseline platelet count and an absence of bleeding. Platelet counts were confirmed on two separate occasions at least 7 days apart when defining complete response or partial response. No response was defined as a platelet count of less than 30×10⁹ cells per L, or less than two-times increase from baseline platelet count, or bleeding.
6-month sustained overall response to ITP treatments | A response lasting for at least 6 months without any additional intervention specific to primary immune thrombocytopenia was defined as a sustained response
  Complete response was defined as a platelet count of 100×10⁹ cells per L or higher and an absence of bleeding. Partial response was defined as a platelet count of 30×10⁹ cells per L or higher, but less than 100×10⁹ cells per L, and at least a doubling of the baseline platelet count and an absence of bleeding. Platelet counts were confirmed on two separate occasions at least 7 days apart when defining complete response or partial response. No response was defined as a platelet count of less than 30×10⁹ cells per L, or less than two-times increase from baseline platelet count, or bleeding.

SECONDARY OUTCOMES:
time to response | an average of 6 months
  the time from treatment initiation to achieve a complete response or a partial response
duration of response | through study completion, an average of one year
  the time from achievement of a complete response or a partial response to the loss of response (platelet count <30×10⁹ cells per L; measured on two occasions more than 1 day apart or the presence of bleeding).
therapy associated adverse events | up to one year
  nausea and diarrhea (report in frequency); pruritus (report in frequency); headache and dizziness (report in frequency)

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hou, MD,PhD, Principal Investigator — Shandong University Qilu Hospital
Locations (2):
- China (2):
  - Qilu hospital, Shandong University, Jinan, Shandong
  - Qilu hospital (Qingdao), Shandong University, Qingdao, Shandong